CLINICAL TRIAL: NCT06927115
Title: Comparative Analysis of Mulligan and Maitland Mobilizations Techniques on Disability and Quality of Life in Adhesive Capsulitis
Brief Title: Comparative Analysis of Mulligan and Maitland Mobilizations Techniques in Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-01005 Rafi Ullah
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Adhesive Capsulitis of Shoulder
Keywords: Adhesive capsulitis; Shoulder joint mobility; Shoulder stiffness
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maitland Mobilization (Experimental): This group will be treated with Maitland mobilization with 30 repetition and 3 set in each repetition 3 time a week for 4 weeks along with conventional exercises like Monkey bar, towel stretching, and codmen exercise.
  Interventions: Other: Maitland Mobilization
- Mulligan Mobilization (Experimental): This group will be treated with Maitland mobilization of the shoulder joint with 30 repetition and 3 set in each repetition 3 time a week for 4 weeks along with conventional exercises like Monkey bar, towel stretching, and codmen exercise.
  Interventions: Other: Mulligan Mobilization

INTERVENTIONS:
Other: Maitland Mobilization — Provide maitland mobilization technique along with conventional exercises like Monkey bar, towel stretching, and codmen exercise to each subject.
  Arms: Maitland Mobilization
Other: Mulligan Mobilization — Provide mulligan mobilization technique along with conventional exercises like Monkey bar, towel stretching, and codmen exercise to each subject.
  Arms: Mulligan Mobilization

SUMMARY:
Mobilization techniques are widely used in physiotherapy to address the pain and stiffness associated with adhesive capsulitis. Two commonly employed approaches are Mulligan's mobilization and Maitland's mobilization, both of which aim to restore joint mobility and improve functional outcomes. However, the relative effectiveness of these techniques in improving disability and quality of life in patients with adhesive capsulitis has not been conclusively established. This study will help to find out the best mobilization option for adhesive capsulitis or frozen shoulder for all four stages of adhesive capsulitis.

DETAILED DESCRIPTION:
Adhesive capsulitis is a condition characterized by pain, loss of both active and passive range motion of the shoulder joint in all planes especially abduction and external rotation. In general population the prevalence of adhesive capsulitis is 2-5% and its incidence is 2%.The prevalence of adhesive capsulitis in diabetic patient is 11- 30% while in non-diabetic is 2-10%.Adhesive capsulitis is more common in women aged between 40-60 years (12). Adhesive capsulitis is bilateral in 20-30 % of cases and the opponent shoulder become involved within five years Based on etiology Adhesive capsulitis is classified into primary or true frozen shoulder and secondary, in primary adhesive capsulitis there is global capsular inflammation without any known cause or pre-existing condition while secondary adhesive capsulitis is associated with any recognized systemic, intrinsic or extrinsic cause. The systemic causes of secondary adhesive capsulitis comprise thyroid diseases, diabetes mellitus and decreased level of adrenaline. The intrinsic cause of secondary adhesive capsulitis is rotator cuff disease andcalcification of tendon or tendonitis. The extrinsic causes of secondary adhesive capsulitis include breast surgery in women, post trauma, clavicle or humerus fracture and early history of cerebral vascular accident

ELIGIBILITY:
Inclusion Criteria:

* Age 35-50 years.
* Diagnosed case of primary adhesive capsulitis.
* Pain and limited range of motion in the affected shoulder. (External rotation>abduction>internal rotation)
* Willing to participate in the study

Exclusion Criteria:

* Previous shoulder surgery.
* Severe osteoporosis or fractures.
* Neurological or rheumatological conditions.
* Neck and cardiac surgery
* History of recent fractures

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
NPRS | six weeks
  The Numeric Pain Rating Scale (NPRS) is a 0 to 10 self-reported scale used to assess pain intensity, where 0 = no pain and 10 = worst possible pain. It is a simple, reliable tool commonly used in clinical trials to measure pain levels before and after interventions.
Goniometer | Six weeks
  A goniometer is a standardized tool used to measure shoulder range of motion (ROM) in degrees. It consists of a protractor with two arms, one stationary and one movable, to assess joint angles during movement.
SPADI | Six weeks
  The Shoulder Pain and Disability Index (SPADI) is a self-reported questionnaire used to assess pain and functional disability in individuals with shoulder conditions. It consists of 13 items divided into two subscales: pain (5 items) and disability (8 items), scored on a 0-100 scale, with higher scores indicating greater impairment
SF- 36 Scale | Six weeks
  The Short Form-36 (SF-36) Health Survey is a validated questionnaire used to assess health-related quality of life (HRQoL) across eight domains, including physical functioning, pain, and general health. It generates physical and mental health summary scores on a 0-100 scale, with higher scores indicating better well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Zavata Afnan, MS NMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University Malakand Campus, Chakdara, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No